CLINICAL TRIAL: NCT00314587
Title: Treatment of Unstable Both-Bone Midshaft Forearm Fractures in Children: A Randomized Trial Between 1 and 2 Elastic Stable Intramedullary Nails
Brief Title: Treatment of Unstable Both-Bone Midshaft Forearm Fractures in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Colaris, Joost, M.D. (Individual)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: colaris01
Record Dates: First submitted 2006-04-12; First posted 2006-04-14 (Estimated); Last update posted 2007-02-26 (Estimated); Status verified 2006-11

CONDITIONS: Fracture
Keywords: fracture; forearm; midshaft; child; treatment
MeSH Terms: conditions — Fractures, Bone

INTERVENTIONS:
Procedure: 1 or 2 elastic stable intramedullary nails

SUMMARY:
The investigators created a randomized clinical trial between 1 or 2 elastic stable intramedullary nails to find out what kind of treatment is optimal for unstable both-bone midshaft forearm fractures.

DETAILED DESCRIPTION:
Children who arrive at the emergency unit with an unstable both-bone midshaft forearm fracture will be asked to join the trial.

If the fracture will be unstable during reposition in the operating room, a randomization between 1 or 2 ESIN will be done.

The aftertreatment will be the same for both groups: above elbow plaster for 3 weeks. Outpatient clinic visits till a follow-up of 9 months. During these visits we will investigate: consolidation and dislocation on X-ray, function of both arms, complaints in daily living and complications.

ELIGIBILITY:
Inclusion Criteria:

* Stable both-bone forearm fracture
* Age < 16 years old
* Dislocation
* Unstable

Exclusion Criteria:

* Fracture older than 1 week
* No informed consent
* Refracture
* Open fracture (Gustillo 2 and 3)

Max Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60
Dates: Start 2006-01

PRIMARY OUTCOMES:
pronation and supination

SECONDARY OUTCOMES:
complications, function, esthetics, complaints in daily living, X-rays

CONTACTS AND LOCATIONS:
Overall Officials: Joost W Colaris, M.D., Principal Investigator — HAGA/Erasmus Medical Centre
Locations (2):
- Netherlands (2):
  - Erasmus Medical Centre, Sophia Children's Hospital, Rotterdam, South Holland
  - HAGA, Juliana Children's Hospital, The Hague, South Holland